CLINICAL TRIAL: NCT03818841
Title: High-flow Nasal Cannula Therapy in the Treatment of Acute Carbon Monoxide Poisoning
Brief Title: The Role of High-flow Nasal Cannula Therapy in the Treatment of Acute Carbon Monoxide Poisoning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-HFNC
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula group (Experimental): Patients randomised in this group will receive oxygen therapy via a high-flow nasal cannula device with a 60 L/min flow and a 100% fraction of inspired oxygen
  Interventions: Device: High-flow nasal cannula device
- Non-rebreathing oxygen mask group (Other): In this group patients will be treated with standard oxygen therapy delivered through a non-rebreathing face mask with a 15 L/min flow
  Interventions: Device: Non-rebreathing oxygen mask group

INTERVENTIONS:
Device: High-flow nasal cannula device — Patients will be randomly allocated to this treatment
  Other Names: AIRVO 2, Fisher & Paykel Healthcare LTD
  Arms: High-flow nasal cannula group
Device: Non-rebreathing oxygen mask group — Patients will be randomly allocated to this treatment
  Other Names: Standard non-rebreathing oxygen mask
  Arms: Non-rebreathing oxygen mask group

SUMMARY:
The aim of the study is to test whether oxygen therapy delivered through high-flow nasal cannula devices in patients admitted to the emergency department for acute carbon monoxide poisoning is superior to the non-rebreathing oxygen face mask therapy with a 15 L/minute oxygen flow (currently the first-line therapy), in terms of reduction of carboxyhemoglobin (COHb) concentration and delayed neurological sequelae incidence.

ELIGIBILITY:
Inclusion Criteria:

* Age v 18 years
* Carbon monoxide intoxication as major problem leading to emergency department admission
* Carboxyhemoglobin (COHb) concentration 10% at the time of enrolment

Exclusion Criteria:

* Age < 18 years
* Glasgow coma scale ≤ 13
* Refusal to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
COHb reduction at 90 minutes | 90 minutes
  Patients in the High-flow nasal cannula group and patients in the non-rebreathing oxygen mask group will be compared in terms of COHb reduction at 90 minutes. The hypothesis is that in patients treated with high flow nasal cannula the reduction in COHb at 90 minutes will be significantly different compared to patients treated with non-rebreathing oxygen mask.

SECONDARY OUTCOMES:
Variation in the incidence of delayed neurologic sequelae | 6 weeks
  Patients in the High-flow nasal cannula group and patients in the non-rebreathing oxygen mask group will be compared in terms of incidence and severity of delayed neurologic syndrome.
  At the time of discharge from the emergency department, each enrolled patient will undergo neurocognitive testing.
  Six weeks after discharge, a follow-up visit for each patient will be performed which will include neurocognitive testing and a functional magnetic resonance imaging, in order to determine the presence of delayed neurologic sequelae.
  Patients in the two groups of treatment will be subsequently compared.
Variation in serum lactate concentration | 6 weeks
  Patients in the High-flow nasal cannula group and patients in the non-rebreathing oxygen mask group will be compared in terms of serum lactate variations. In particular, serum lactate levels will be evaluated at different time points, in order to test whether different treatments lead to different kinetic.
Variation in serum troponin concentration | 6 weeks
  Patients in the High-flow nasal cannula group and patients in the non-rebreathing oxygen mask group will be compared in terms of troponin concentration variations. In particular, serum troponin levels will be evaluated at different time points, in order to test whether different treatments lead to different kinetic.
Variation in S100B levels concentration | 6 weeks
  Patients in the High-flow nasal cannula group and patients in the non-rebreathing oxygen mask group will be compared in terms of serum protein S100B variations. In particular, protein S100B will be evaluated at different time points, in order to test whether different treatments lead to different protein kinetic.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi M Castello, MD, Principal Investigator — A.O.U. Maggiore della Carità di Novara
Locations (1):
- AOU Maggiore della Carità di Novara. Emergency Medicine Department. Department of Translational Medicine., Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brotfain E, Zlotnik A, Schwartz A, Frenkel A, Koyfman L, Gruenbaum SE, Klein M. Comparison of the effectiveness of high flow nasal oxygen cannula vs. standard non-rebreather oxygen face mask in post-extubation intensive care unit patients. Isr Med Assoc J. 2014 Nov;16(11):718-22. PMID 25558703
- [Result] Jeon SB, Sohn CH, Seo DW, Oh BJ, Lim KS, Kang DW, Kim WY. Acute Brain Lesions on Magnetic Resonance Imaging and Delayed Neurological Sequelae in Carbon Monoxide Poisoning. JAMA Neurol. 2018 Apr 1;75(4):436-443. doi: 10.1001/jamaneurol.2017.4618. PMID 29379952
- [Result] Rose JJ, Wang L, Xu Q, McTiernan CF, Shiva S, Tejero J, Gladwin MT. Carbon Monoxide Poisoning: Pathogenesis, Management, and Future Directions of Therapy. Am J Respir Crit Care Med. 2017 Mar 1;195(5):596-606. doi: 10.1164/rccm.201606-1275CI. PMID 27753502
- [Result] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645